CLINICAL TRIAL: NCT04766164
Title: Health Beliefs, Behaviors, and Healthcare Experiences Among a National Sample of United States Young and Mid-Age Adults
Brief Title: Health Beliefs, Behaviors, and Healthcare Experiences Among United States Young and Mid-Age Adults
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-20853
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: HPV Vaccine Knowledge
Keywords: HPV; HPV Vaccine
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Males and Females ages 18-26: Participants between the ages of 18-26 will complete a survey
  Interventions: Behavioral: Survey
- Males and Females ages 27-45: Participants between the ages of 27-45 will complete a survey
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Data will be obtained via self-report from participants via a one-time Qualtrics survey.

SUMMARY:
The study will provide important insight into current HPV vaccine knowledge/awareness, health beliefs, affect, vaccine discussions, decision preparedness, and vaccine intentions and behaviors among those ages 18-45, while examining potential differences in responses between those ages 18-26 and those ages 27-45 and vaccinated and unvaccinated individuals.

DETAILED DESCRIPTION:
The study will provide important insight into current HPV vaccine knowledge/awareness, health beliefs, affect, vaccine discussions, decision preparedness, and vaccine intentions and behaviors among those ages 18-45, while examining potential differences in responses between those ages 18-26 and those ages 27-45 and vaccinated and unvaccinated individuals. In addition, the study will illuminate gaps in knowledge and awareness as well as the education intervention preferences (e.g., intervention platform, source of information, timing of intervention) of individuals ages 18-45. Among those ages 27-45, shared clinical decision-making is recommended. Compared to individuals ages 18-26, individuals ages 27-45 may need to be supported uniquely so that they are prepared to engage in shared clinical decision-making about HPV vaccination with their healthcare provider. Thus, among unvaccinated individuals ages 27-45, for whom shared clinical decision-making is recommended, preparedness for engagement in shared clinical decision-making will be assessed and explored. The study also will allow investigators to identify how best to target information to young adults and mid-adults both for themselves, and among those with children, for their children.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Living in the United States
* a KnowledgePanel panelist directly or via verified partners
* Have internet access
* Able to read, write and understand English
* Individuals can participant regardless of their HPV vaccination status

Exclusion Criteria:

* Individuals who do not meet inclusion criteria

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Participants living throughout the United States
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
HPV Vaccine Knowledge | Day 1
  Data from survey will describe HPV and HPV vaccine knowledge, health beliefs, attitudes, affect, health literacy, health care experiences, vaccine discussions and information sources, preparedness for shared decision-making and HPV vaccine uptake and intentions and examine relationships between these variables among a national sample of U.S. adults (N=4,000) ages 18-45 years.
HPV-Related Educational Intervention Preferences | Day 1
  Data from survey will describe intervention preferences and associations between intervention preferences and sociodemographic variables (e.g., age, gender, race, ethnicity, socioeconomic status, employment status, parental status, and insurance status).

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Christy, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States